CLINICAL TRIAL: NCT00386828
Title: Phase II Study of Chemoradiation for Locally Advanced and Low Rectal Cancers: Avastin-Capecitabine-Oxaliplatin-Radiation REctal Cancer Trial
Brief Title: Chemoradiation for Locally Advanced and Low Rectal Cancers: Avastin-Capecitabine-Oxaliplatin-Radiation REctal Cancer Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Dr Hagen Kennecke, BC Cancer Agency - Vancouver Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROTOCOL NUMBER: OZM-004; A-CORRECT Study
Record Dates: First submitted 2006-10-11; First posted 2006-10-12 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Advanced Colorectal Cancer
Keywords: colorectal cancer; advanced colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bevacizumab:

SUMMARY:
This phase II study will evaluate the effect of bevacizumab, capecitabine and oxaliplatin with radiation on rectal cancer. Researchers will also evaluate the tolerability (how it makes the patient feel) and safety of this combination by watching for harmful side-effects.It is hoped that by adding bevacizumab to the capecitabine/oxaliplatin treatment in combination with radiation before surgery will improve response rate.

DETAILED DESCRIPTION:
Improved pre-operative therapy is required in the management of high risk rectal cancer in order to decrease local recurrence and increase the rate of sphincter sparing surgery. Capecitabine, oxaliplatin and bevacizumab represent new systemic agents and have been given safely in phase I and II trials concurrently with radiation with promising improvements in pCR rates of 15 -24% compared to historic rates of 8-14% achieved with 5-FU alone. Improvements in pCR rates have not been associated with an increase in post-operative complication rates. A trial of all three of these agents is justified due to their enhanced efficacy when given in combination as well as their non-overlapping treatment toxicity profile.

This is a one-armed, multi-centred, Phase II study in patients with T3/4 locally advanced and T3/4 low lying rectal cancer, to study the efficacy and safety of the addition of bevacizumab to a regimen of capecitabine and oxaliplatin in combination with pre-operative radiation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the rectum, defined as either:

Mid- or upper rectal tumours (>= 6 - 15 cm): T3 or T4 adenocarcinoma that is fixed or partially fixed or tethered and is potentially resectable; or Low rectal tumours (<6cm): T3 or T4 adenocarcinoma: or Node positive rectal tumours (<= 15cm): T1-4N2 or T1-4N+ where pelvic nodes approach or invade the mesorectum.

M0/X or M1 is permitted as long as definitive resection of the primary tumour is planned and, in the opinion of the investigator, it is safe to delay full dose of systemic chemotherapy

* Appropriate staging investigations of the primary tumour, either endorectal ultrasound or pelvic MRI.
* Male or female aged 18 or older.
* Have a performance status ECOG of 0 or 1.
* Have a life expectancy greater than 6 months.
* Adequate organ function and coagulation parameters as measured by:

ANC >=1.5 platelets >=100 Serum creatinine <= 1.5X ULN AST, ALT <= 2.5X ULN Bilirubin <= 1.5 ULN PTT and INR within normal limits Albumin >= than 30

* Patient consent
* No neurological diseases that can increase the neurotoxicity of oxaliplatin
* Be willing and able to comply with the protocol for the duration of the study.

Exclusion Criteria:

* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day -14, (i.e. patients must have recovered from any major surgery), or anticipation of need for major surgical procedure during or within 7 weeks after chemo-radiotherapy.
* Known to have clinical or radiological evidence of CNS metastases.
* Patients with a past or current history (within last 2 years) of other malignancies, except for the indication under this study and curatively treated basal and squamous skin cancer or in-situ cancer of the cervix.
* Women of childbearing potential with either a positive or no pregnancy test at baseline or lactating. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study. Patients of childbearing potential must be willing to use a reliable method of birth control. i.e.: doublebarrier method, oral contraceptive, implant, dermal contraception, long-term injectable contraceptive, intrauterine device or tubal ligation during the study
* Evidence of bleeding diathesis or coagulopathy.
* Uncontrolled hypertension, defined as SBP > 150/100 on more than one occasion that does not respond to therapy with antihypertensive agents
* Clinically significant (i.e. active) cardiovascular disease for example:

cerebrovascular accidents (<=6 months), myocardial infarction (<= 6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication.

* Current or recent (within 10 days prior to study treatment start) ongoing treatment with anticoagulants for therapeutic purposes i.e. except for anticoagulation for maintenance of patency of permanent indwelling IV catheters.
* Evidence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or puts the patient at high risk from treatment complications.
* Ongoing treatment with aspirin (> 325 mg/day) or other medications known to predispose to gastrointestinal ulceration.
* Any other serious or uncontrolled illnesses.
* Current or recent serious polyneuropathy.
* Known hypersensitivity against bevacizumab.
* Known peripheral neuropathy >= NCI CTCAE grade 1. Absence of deep tendon reflexes (DTRs) as the sole neurologic abnormality does not render the patient ineligible.
* Organ allografts requiring immunosuppressive therapy.
* Serious, non-healing wound, ulcer, or bone fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is pathologic complete response (pCR) rate

SECONDARY OUTCOMES:
Rate of Sphincter Sparing Surgery:
Complete Resection Rate
Post-Surgical Complication Rates:

CONTACTS AND LOCATIONS:
Overall Officials: Hagen Kennecke, MD, Study Chair — BC Cancer Agency -Vancouver Centre
Locations (6):
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Centre for Southern Interior, Kelowna, British Columbia
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario